CLINICAL TRIAL: NCT03315949
Title: Comparison of Bowel Cleansing Efficacy Between Same-day Dose Versus Split Dose : A Single Center, Operator Blinded, Prospective Randomized Controlled Trial
Brief Title: Comparison of Bowel Cleansing Efficacy Between Same-day Dose Versus Split Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Tae-Geun Gweon, Clinical associate professor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OC17MESI0060
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Unrecognized Condition
MeSH Terms: interventions — Polyethylene Glycols; Golytely

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Same-day dose group (Experimental): Participants who ingest bowel cleanser on the day of colonoscopy. Participant will ingest the 4L PEG on the day of colonoscopy.
  Interventions: Drug: Polyethylene Glycol (PEG)
- Split-dose group (Active Comparator): Participants who ingest bowel cleanser by split dose. 2L PEG will be ingested 1 day before colonoscopy. Remaining 2L bowel cleanser will be ingested on the day of colonoscopy.
  Interventions: Drug: Polyethylene Glycol (PEG)

INTERVENTIONS:
Drug: Polyethylene Glycol (PEG) — Different method for bowel cleansing using same bowel cleanser. Same-day dose group : 4L PEG will be ingested on the day of colonoscopy Spli-dose group : 2L PEG will be ingested 1 day before colonoscopy, remaining 2L PEG will be ingested on the day of colonoscopy
  Other Names: colyte

SUMMARY:
Split dose bowel cleansing is recommended method for colonoscopy. For afternoon colonoscopy, same-day dose of bowel cleansing is alternative option. Recently, same-day bowel cleansing for morning colonoscopy was validated. To date, there was no study which compared the bowel cleansing efficacy between same-day dose and split dose regardless of colonoscopy time. The aim of current study is to compare the bowel cleansing efficacy, adverse events, and patient's tolerability between the two group.

Subjects who underwent colonoscopy for various reasons were included. After agreeing to participate in the study, study participants were randomly assigned to split dose or same day dose group. Bowel cleansing is done using polyethylene glycol (PEG). All colonoscopy was done between 10 AM to 6 PM. Study participants were instructed to ingest 500ml PEG every 15 minutes. Subjects who were assigned to split dose group ingested 2L PEG from 9PM 1 day before colonoscopy. Remaining 2L PEG was ingested 3-5 hours before colonoscopy. In the same-day dose group, bowel cleansing was started from 5AM for subjects who were scheduled to receive colonoscopy in the morning. Afternoon colonoscopy group in the same-day dose group ingested 2L PEG from 5AM. Remaining 2L PEG was finished 3-5 hours before colonoscopy.

Bowel cleansing efficacy was assessed using Boston bowel preparation scale. Vital signs and laboratory tests were checked before colonoscopy. Study participants completed questionnaire which contained patient's satisfaction, tolerability, and adverse event during bowel cleansing. Bowel cleansing efficacy, patient's tolerability, and safety profile were compared between the two groups. Successful bowel cleansing was estimated 85% for split dose group.

The investigators set 10% for inferior margin. Considering 10% drop out, a total of 352 subjects will be recruited.

DETAILED DESCRIPTION:
Randomization and blinding:

Randomization will be done using computer generated randomization list. A specialized nurse will explain the method of bowel cleansing. Investigators (endoscopists) are blinded to bowel cleansing method.

Endpoint:

Primary end point is successful bowel cleansing rated by Boston bowel preparation (BBPS) scale. Successful bowel cleansing is defined as all segment is 2 or 3 points. Endoscopists will assess BBPS when colonoscopy withdrawal.

Secondary end point was patient's tolerability and safety profile including adverse events. Patient's satisfaction to the different bowel cleansing method and adverse events (nausea, vomiting, dizziness, fatigue) will be investigated by questionnaire before colonoscopy. Blood test will be done before colonoscopy.

Statistical analysis:

Bowel cleansing success, patient's tolerability and safety profile will be compared between the two groups. Student t test for continuous variables and the chi-square test or Fisher exact test for categorical variables.

Sample size:

This study is non-inferioty study. Assuming bowel cleansing success rate 85% in the split-dose group, the significant difference between the two groups were hypothesized at 10%. Considering 80% power and 10% drop rate, a total of 352 participants is needed.

ELIGIBILITY:
Inclusion Criteria:

* all subjects who undergo colonoscopy for various reasons.

Exclusion Criteria:

* hemodynamic instability
* ileus or bowel obstruction
* active inflammatory bowel disease
* advanced colon cancer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Geun Gweon, Ph.D, Principal Investigator — Professor
Locations (1):
- Incheon St. Mary's Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Same-day Dose Group: Participants who ingest bowel cleanser on the day of colonoscopy. Participant will ingest the 4L PEG on the day of colonoscopy.
  Polyethylene Glycol (PEG): Different method for bowel cleansing using same bowel cleanser.
  Same-day dose group : 4L PEG will be ingested on the day of colonoscopy Spli-dose group : 2L PEG will be ingested 1 day before colonoscopy, remaining 2L PEG will be ingested on the day of colonoscopy
- Split-dose Group: Participants who ingest bowel cleanser by split dose. 2L PEG will be ingested 1 day before colonoscopy. Remaining 2L bowel cleanser will be ingested on the day of colonoscopy.
  Polyethylene Glycol (PEG): Different method for bowel cleansing using same bowel cleanser.
  Same-day dose group : 4L PEG will be ingested on the day of colonoscopy Spli-dose group : 2L PEG will be ingested 1 day before colonoscopy, remaining 2L PEG will be ingested on the day of colonoscopy
Period: Overall Study
Arm/Group | Same-day Dose Group | Split-dose Group
Started | 176 | 176
Completed | 171 | 166
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Population: Participants who ingested bowel cleansing agent according to protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Same-day Dose Group | Split-dose Group | Total
Number analyzed (Participants) | 172 | 167 | 339
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 122 | 244
  >=65 years | 50 | 45 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (8.5) | 58.4 (9.4) | 58.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 72 | 144
  Male | 100 | 95 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 172 | 167 | 339
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 172 | 167 | 339

OUTCOME MEASURES:

1. Primary Outcome: Boston Bowel Preparation Scale
Description: Primary endpoint=Successful bowel cleansing (all segmental score 2 or above)
  * Boston bowel preparation scale (0-9) Sum of 3 segment of bowel. 0=inadequate
  1. poor
  2. good
  3. excellent
Time Frame: Bowel cleansing efficacy using Boston bowel preparation scale will be assessed during colonoscopy withdrawal
Measure: Number; unit: Number of successful cleansing
Arm/Group | Same-day Dose Group | Split-dose Group
Number analyzed (Participants) | 171 | 166
Number of successful cleansing | 169 | 163

ADVERSE EVENTS:
Time Frame: Adverse events were collected between enrollment and 4 weeks of procedure
Arm/Group | Same-day Dose Group | Split-dose Group
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/167
Serious Adverse Events (participants affected / at risk) | 0/172 | 0/167
Other Adverse Events (participants affected / at risk) | 73/172 | 67/167
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Same-day Dose Group (N=172) | Split-dose Group (N=167)
Adverse events related to bowel cleanser (Gastrointestinal disorders) | 41 (41) | 33 (33) — nausea
Adverse events related to bowel cleansing agent (Gastrointestinal disorders) | 23 (23) | 13 (13) — vomiting
Adverse events related to bowel cleansing agent (Gastrointestinal disorders) | 16 (16) | 20 (20) — bloating
Adverse events related to bowel cleansing agent (Nervous system disorders) | 8 (8) | 9 (9) — Headache, dizziness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT03315949/Prot_SAP_000.pdf